CLINICAL TRIAL: NCT01757171
Title: An Open-Labeled, Multicenter Phase II Study of Cabazitaxel in Refractory Metastatic Gastric or Gastroesophageal Adenocarcinoma
Brief Title: Phase II Study of Cabazitaxel in Refractory Metastatic Gastric or Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208012946
Record Dates: First submitted 2012-12-06; First posted 2012-12-28 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Adenocarcinoma; Distal Esophageal Adenocarcinoma
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (taxane naïve) (Experimental): No prior Taxane treatment. Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks
  Interventions: Drug: Cabazitaxel
- Arm B (prior taxane therapy) (Experimental): Subject previously treated with taxane. Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 20mg IV over 1 hour every 3 weeks

SUMMARY:
Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks, as is the standard administration dose and schedule. This application is a non-labeled indication for cabazitaxel and will inform future drug development in gastroesophageal malignancies, where docetaxel remains an approved first line agent, but is not routinely used due to excessive toxicity and marginal efficacy.

At the conclusion of this study, we hope to demonstrate activity of single agent cabazitaxel in refractory gastric cancer, with preferential activity in one or more gastric cancer subtypes

DETAILED DESCRIPTION:
Prior to initiating protocol therapy, patients will undergo screening evaluations, to be done within 30 days of protocol initiation unless otherwise noted.

Patients who are taxane naïve will be assigned to arm A and patients who have had prior taxane therapy will be assigned to Arm B. Each arm will be analyzed separately for the primary study endpoint of 3 month progression free survival rate (PFS), as defined as the time from the start of treatment to the date of disease progression or death. Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks.

In the absence of treatment delays due to adverse event(s), treatment may continue until disease progression; intercurrent illness that prevents further administration of treatment; unacceptable adverse event(s); patient decides to withdraw; general or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

Patients will be followed for 6 months after removal from study or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have histologically or cytologically confirmed gastric, or gastroesophageal adenocarcinoma, or distal esophageal adenocarcinoma.
2. Subject must have unresectable or metastatic gastroesophageal adenocarcinoma.
3. Subject must have evaluable disease as per RECIST criteria.
4. Subject must have had at least one prior cytotoxic chemotherapy regimen for unresectable or metastatic disease. Prior taxane therapy is allowed.
5. Age >/=18 years old.
6. ECOG performance status status >/= 2
7. Subject must have normal organ and marrow function as defined below:

   * WBC >/= 3,000/uL
   * Total Bilirubin ≤ 1.5 x upper limits of normal
   * AST (SGOT) ≤ 2.5 x upper limits of normal
   * ALT (SGPT) ≤ 2.5 x upper limits of normal
   * Hgb > 7.5 g/dl (without transfusion within 7 days)
   * ANC > 1000 /ml
   * Plt > 75 K/ml (without transfusion)
   * Creatinine* < 2.0 g/dl *or a calculated creatinine clearance > 45/cc (using Cockroft-Gault formula)

9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. 10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subject with previously untreated unresectable or metastatic gastroesophageal adenocarcinoma.
2. Subject with more than 2 prior cytotoxic therapies (not including treatment administered for locally curable disease) for unresectable or metastatic gastroesophageal adenocarcinoma.
3. Subject with CNS metastases with active neurologic dysfunction. These patients are excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse event.
4. Significant medical co-morbidity that would preclude safe administration of cytotoxic therapy, including but not limited to:

   a.Cardiac disease i. Unstable angina ii. Myocardial infarction < 3 months prior to study initiation b. Ongoing serious infection i. Bacteremia or sepsis requiring intravenous antibiotics ii. HIV with AIDS defining illness c.Inadequate oral nutritional intake i. Requirement for daily intravenous fluids or total parenteral nutrition. d. Psychiatric illness/social situations that would limit compliance with study requirement
5. Subject who has had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from prior treatment related toxicity with persistent symptoms >/= grade 2 due to agents administered more than 4 weeks earlier.
6. Subject may not receive another investigational agent.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cabazitaxel, or to drugs formulated with polysorbate 80.
8. Pregnant (positive pregnancy test) and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (5):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Taxane naïve): Arm A - No prior Taxane treatment. Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks Cabazitaxel: 20mg IV over 1 hour every 3 weeks
- Arm B (Prior Taxane Therapy): Arm B - Subject previously treated with taxane. Cabazitaxel will be administered 20 mg/m2 IV over 1 hour every 3 weeks Cabazitaxel: 20mg IV over 1 hour every 3 weeks
Period: Overall Study
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Started | 61 | 24
Completed | 53 | 23
Not Completed | 8 | 1
Not completed — Adverse Event | 5 | 1
Not completed — Disease Progression | 1 | 0
Not completed — Hospitalization | 1 | 0
Not completed — ECOG decline | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy) | Total
Number analyzed (Participants) | 53 | 23 | 76
Age, Continuous [Median (Full Range); unit: years] | 62.1 [35.46 to 91.76] | 57.34 [36.89 to 73.45] | 61.67 [35.46 to 91.76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 6 | 26
  Male | 33 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 36 | 14 | 50
  Unknown or Not Reported | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 36 | 14 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 23 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression at the 3 Month Follow up Visit
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions Results below list the number of participants who progressed at the 3 month follow up visit
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Number analyzed (Participants) | 53 | 23
participants | 15 | 7

2. Secondary Outcome: Duration of Event Free Survival of Subjects Treated With Cabazitaxel
Description: To examine other measures of efficacy such as overall progression free in all evaluable patients
Time Frame: From date of first subject treated until the date of last subject documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Number analyzed (Participants) | 53 | 23
months | 2.17 [1.31 to 2.6] | 1.31 [1.15 to 3.98]

3. Secondary Outcome: Number of Participants With Response to Cabazitaxel Across Gastric Cancer Subtypes
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Number analyzed (Participants) | 53 | 22
participants
  Stable Disease | 12 | 5
  Partial Response | 5 | 3
  Complete Response | 1 | 0
  Progression Disease | 34 | 14
  Death | 1 | 0

4. Secondary Outcome: Percent of Participants Treated With Cabazitaxel With Event Free Survival
Description: To examine other measures of efficacy such as overall survival in all evaluable patients
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Number analyzed (Participants) | 53 | 23
percentage of participants | 11.32 [4 to 23] | 13 [3 to 34]

ADVERSE EVENTS:
Arm/Group | Arm A (Taxane naïve) | Arm B (Prior Taxane Therapy)
Serious Adverse Events (participants affected / at risk) | 27/53 | 15/23
Other Adverse Events (participants affected / at risk) | 53/53 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Taxane naïve) (N=53) | Arm B (Prior Taxane Therapy) (N=23)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Acute Kidney Failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Decreased white blood cell count (Investigations) | 4 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heart Block (Cardiac disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (General disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Increased generalized weakness (General disorders) | 1 (1) | 1 (1)
Nausea (General disorders) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 6 (6) | 8 (9)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Right Upper Quadrant Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Taxane naïve) (N=53) | Arm B (Prior Taxane Therapy) (N=27)
Anemia (Blood and lymphatic system disorders) | 25 (34) | 13 (19)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leuocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left Neck Adenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Epistaxis (nose bleeds) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Complete heart block (Cardiac disorders) | 1 (1) | 0 (0)
Heart Disease (Organic) (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
sound in ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
erythema at the bottom of eyelids (Eye disorders) | 1 (1) | 0 (0)
increased tears (Eye disorders) | 0 (0) | 1 (1)
vision change (Eye disorders) | 1 (1) | 0 (0)
Right eye Pressure (Eye disorders) | 1 (1) | 0 (0)
right eye dimness (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 25 (27) | 9 (13)
Ascites (Gastrointestinal disorders) | 6 (6) | 5 (6)
Bloating (Gastrointestinal disorders) | 7 (7) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (20) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 14 (20) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 13 (16) | 2 (3)
Esophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (9) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (3) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 24 (31) | 12 (16)
Rectal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (18) | 9 (13)
Increased Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in anterior ribs (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia (Gastrointestinal disorders) | 2 (3) | 0 (0)
mouth sore (Gastrointestinal disorders) | 1 (1) | 1 (1)
hiatus hernia syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increasing Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
early satiety (Gastrointestinal disorders) | 1 (1) | 0 (0)
difficulty swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0)
pyloric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
early satiety (Gastrointestinal disorders) | 1 (1) | 1 (1)
left upper quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
extensive peritoneal carcinomatosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
H.Pylori Infection (Gastrointestinal disorders) | 2 (2) | 0 (0)
increase sputum production (Gastrointestinal disorders) | 1 (1) | 0 (0)
bloody stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercholesterolemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melena (black feces) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
epigastralgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral thrush (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anasarca (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clostridium difficle (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased Abdominal Girth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Right Upper Quadrant Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
burping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (Gastrointestinal disorders) | 9 (11) | 1 (1)
Edema limbs (Gastrointestinal disorders) | 9 (11) | 7 (7)
Fatigue (Gastrointestinal disorders) | 47 (64) | 19 (26)
Fever (Gastrointestinal disorders) | 4 (5) | 2 (3)
Localized edema (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malaise (Gastrointestinal disorders) | 4 (4) | 1 (1)
Non-cardiac chest pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rigors (Gastrointestinal disorders) | 0 (0) | 1 (1)
Big white light and dizziness (Gastrointestinal disorders) | 0 (0) | 1 (1)
intermittent low appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lightheadedness (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weakness (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema- Scrotal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash on Neck (Gastrointestinal disorders) | 0 (0) | 1 (1)
neuropathy to fingers (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight Change (Gastrointestinal disorders) | 2 (2) | 1 (1)
Skin Changes (Gastrointestinal disorders) | 0 (0) | 1 (1)
Body aches (Gastrointestinal disorders) | 0 (0) | 1 (1)
hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypokalemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated CEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
cold intolerance (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion related reaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion site extravasation (Gastrointestinal disorders) | 1 (1) | 0 (0)
uremia (Gastrointestinal disorders) | 1 (1) | 0 (0)
dehydration (Gastrointestinal disorders) | 1 (2) | 0 (0)
Itching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abrasion on R forearm after CT Scan (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (4) | 0 (0)
hypersensitivity to oxaliplatin (Gastrointestinal disorders) | 1 (1) | 0 (0)
vasogenic edema (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLE Edema (Gastrointestinal disorders) | 1 (1) | 0 (0)
moon face (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypocalcemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIGH ALKALINE PHOSPHATASE (Gastrointestinal disorders) | 3 (4) | 0 (0)
HYPOALBUMINEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
general discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neuropathy to Extremities (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cold (Gastrointestinal disorders) | 2 (3) | 0 (0)
Swelling from Contrast Dye (Gastrointestinal disorders) | 1 (1) | 0 (0)
Discharge from Feeding Tube (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
biopsy site sore and numb (Gastrointestinal disorders) | 1 (1) | 0 (0)
Night Sweats (Gastrointestinal disorders) | 1 (2) | 0 (0)
arthralgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
myalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrush (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevate Liver Functions (Hepatobiliary disorders) | 1 (1) | 0 (0)
Splenic Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
mild jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Allergy to Penecillin (Immune system disorders) | 1 (1) | 0 (0)
flu (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Mycoplasma pneumoniae (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter baumanii bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Positive blood culture (Infections and infestations) | 0 (0) | 1 (1)
Bacteruria (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Pain (left side) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
decreseaed neutrophill count (Investigations) | 3 (4) | 3 (4)
Elevated ANC (Investigations) | 1 (1) | 0 (0)
decreased absolute lymphocyte count (Investigations) | 0 (0) | 1 (1)
decreased platelets (Investigations) | 5 (8) | 1 (2)
decreased WBC count (Investigations) | 9 (14) | 7 (10)
Weight gain (Investigations) | 9 (10) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Early Satiety (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dysguesia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Poor Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Poor Oral Intake (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
vitamin B12 defeciency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron defeciency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D3 defeciency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesteremias (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Difficulty Feeding (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspepsia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
right upper quadrant pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower extremity chills at night (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
bone metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
shallow white-based ulcer on L Lower buccal mucosa near border of lip (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
new left cervical and supraclavicular adenopathy of the axilla (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone Mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Dysgeusia (Nervous system disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (3)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (2)
balance difficulty (Nervous system disorders) | 0 (0) | 1 (1)
generalized weakness (Nervous system disorders) | 0 (0) | 2 (2)
hypersensitivity (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 5 (8) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (20) | 7 (9)
reduced dexterity (right hand) (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
brain metastases (Nervous system disorders) | 1 (1) | 0 (0)
right arm spasms (Nervous system disorders) | 1 (1) | 0 (0)
TINGLING IN HANDS (Nervous system disorders) | 1 (1) | 0 (0)
vocal chord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 14 (14) | 5 (5)
Depression (Psychiatric disorders) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (8) | 5 (6)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 1 (1) | 0 (0)
night sweats (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 12 (18) | 2 (4)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (5)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1)
overactive bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
UROSEPSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
left ureteral stricture (Renal and urinary disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
decreased urine output (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (4) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (6) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bengin enlargement of Prostate (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Kidney Stone) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydrouretroneprosis (Renal and urinary disorders) | 0 (0) | 1 (1)
benign prostatic hypertrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Difficulty Urinating (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Renal and urinary disorders) | 0 (0) | 1 (1)
increase in size of right testis (Renal and urinary disorders) | 1 (1) | 0 (0)
post menopausal vaginal bleeding (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0)
Aspiration (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Renal and urinary disorders) | 6 (8) | 4 (4)
Dyspnea (Renal and urinary disorders) | 11 (13) | 6 (9)
Hiccups (Renal and urinary disorders) | 3 (3) | 1 (1)
Hoarseness (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypoxia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Renal and urinary disorders) | 1 (1) | 0 (0)
rales at the bases (Renal and urinary disorders) | 1 (1) | 0 (0)
COPD exacerbation (Renal and urinary disorders) | 1 (1) | 0 (0)
increase mucus production (Renal and urinary disorders) | 1 (1) | 0 (0)
increased mucus (Renal and urinary disorders) | 1 (1) | 0 (0)
Decreased breathing sounds over Left Lower Lung Field (Renal and urinary disorders) | 1 (1) | 0 (0)
Shortness of Breath (Renal and urinary disorders) | 3 (3) | 0 (0)
Pleural effusion (Renal and urinary disorders) | 2 (2) | 0 (0)
Pneumonitis (Renal and urinary disorders) | 2 (2) | 0 (0)
Postnasal drip (Renal and urinary disorders) | 1 (2) | 0 (0)
Sleep apnea (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nasal congestion (Renal and urinary disorders) | 0 (0) | 1 (1)
Shortness of Breath (Renal and urinary disorders) | 0 (0) | 1 (1)
VATS pleurodesis (Renal and urinary disorders) | 0 (0) | 1 (1)
increase in size of right testis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
post menopausal vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VATS pleurodesis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rales at the bases (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
increase mucus production (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decreased breathing sounds over Left Lower Lung Field (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
eczemarous dermatitis with eosinophilic folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritic maculaopapular rash LUQ (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rosacia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills/ Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
psoriasis flare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Puncture Wound Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ecchymotic rash on hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Darkening of skin surrounding nasal areas (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
slow skin turgor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nodular findings (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (7) | 2 (2)
peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0)
scatter petechiae (Vascular disorders) | 1 (1) | 0 (0)
bloody nose (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
portal vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
easy bruisability (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes